CLINICAL TRIAL: NCT05758194
Title: Protective Strategies to Mitigate Post-Operative Right Ventricular (PV) Dysfunction After Centrifugal Flow Durable Left Ventricular Assist Device (LVAD) Implantation
Brief Title: Mitigating Post-Op RV Dysfunction After LVAD Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-0972
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Right Ventricular Dysfunction; Right Ventricular Failure
Keywords: LVAD; LVAD-related complications; right ventricular dysfunction; hemocompatibility-related adverse events; hemodynamic-related events; post-operative right ventricular management; right ventricular failure
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Right

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standardized RV Management (Active Comparator): Physicians will follow prespecified parameters for RV management (consistent with SOC)
  Interventions: Other: Standardized RV Management
- Usual Care RV Management (Active Comparator): Physicians will use their own clinical judgement with no prespecified goals for RV management parameters (consistent with SOC)
  Interventions: Other: Usual Care RV Management

INTERVENTIONS:
Other: Standardized RV Management — Standardized parameters for post-operative management (i.e., Rhythm Management, Ventilation Management, RV Ischemia Management, RV Preload, RV Afterload, RV Contractility, and RV Geometry)
  Arms: Standardized RV Management
Other: Usual Care RV Management — No standardized parameters for post-operative management (i.e., Rhythm Management, Ventilation Management, RV Ischemia Management, RV Preload, RV Afterload, RV Contractility, and RV Geometry)
  Arms: Usual Care RV Management

SUMMARY:
This project evaluates right ventricle (RV) protective strategies after left ventricular assist device (LVAD) implantation.

DETAILED DESCRIPTION:
The main purpose of this study is to learn more about protecting against RV dysfunction and RV failure (RVF) in patients receiving LVAD implantations.

This is a prospective, randomized controlled study that will include 20 patients with heart failure undergoing LVAD implantation. Patients will receive their LVAD implantation as part of routine care. Patients will be randomized 1:1 to one of two arms, 1) standardized RV management arm, and 2) usual care RV management arm, which are both consistent with standard of care (SOC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing durable LVAD implantation without plan for perioperative right ventricular mechanical circulatory support

Exclusion Criteria:

* Patients with pre-operative right ventricular mechanical circulatory support or having high likelihood of requiring right ventricular mechanical circulatory support.
* Patients with RV implantable cardiac device (ICD)/pacemaker lead who are pacemaker-dependent
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Change in right atrial pressure (RAP) pre-LVAD implantation to post-operative day 3 | Baseline, Day 3
  RAP measured by pulmonary artery catheter
Change in right atrial pressure (RAP) pre-LVAD implantation to post-operative day 7 | Baseline, Day 7
  RAP measured by pulmonary artery catheter
Change in right atrial pressure (RAP) pre-LVAD implantation to end of hemodynamic monitoring post-LVAD implantation | Baseline, end of hemodynamic monitoring (about Day 10)
  RAP measured by pulmonary artery catheter
Change in right atrial pressure/pulmonary capillary wedge pressure (RAP/PCWP) pre-LVAD implantation to post-operative day 3 | Baseline, Day 3
  RAP/PCWP measured by pulmonary artery catheter
Change in right atrial pressure/pulmonary capillary wedge pressure (RAP/PCWP) pre-LVAD implantation to post-operative day 7 | Baseline, Day 7
  RAP/PCWP measured by pulmonary artery catheter
Change in right atrial pressure/pulmonary capillary wedge pressure (RAP/PCWP) pre-LVAD implantation to end of hemodynamic monitoring post-LVAD implantation | Baseline, end of hemodynamic monitoring (about Day 10)
  RAP/PCWP measured by pulmonary artery catheter
Change in pulmonary artery pulsatility index (PAPI) pre-LVAD implantation to post-operative day 3 | Baseline, Day 3
  PAPI measured by pulmonary artery catheter
Change in pulmonary artery pulsatility index (PAPI) pre-LVAD implantation to post-operative day 7 | Baseline, Day 7
  PAPI measured by pulmonary artery catheter
Change in pulmonary artery pulsatility index (PAPI) pre-LVAD implantation to end of hemodynamic monitoring post-LVAD implantation | Baseline, end of hemodynamic monitoring (about Day 10)
  PAPI measured by pulmonary artery catheter
Change in right ventricle stroke work index (RVSWI) pre-LVAD implantation to post-operative day 3 | Baseline, Day 3
  RVSWI measured by pulmonary artery catheter
Change in right ventricle stroke work index (RVSWI) pre-LVAD implantation to post-operative day 7 | Baseline, Day 7
  RVSWI measured by pulmonary artery catheter
Change in right ventricle stroke work index (RVSWI) pre-LVAD implantation to end of hemodynamic monitoring post-LVAD implantation | Baseline, end of hemodynamic monitoring (about Day 10)
  RVSWI measured by pulmonary artery catheter
Change in cardiac power output (CPO) pre-LVAD implantation to post-operative day 3 | Baseline, Day 3
  CPO measured by pulmonary artery catheter
Change in cardiac power output (CPO) pre-LVAD implantation to post-operative day 7 | Baseline, Day 7
  CPO measured by pulmonary artery catheter
Change in cardiac power output (CPO) pre-LVAD implantation to end of hemodynamic monitoring post-LVAD implantation | Baseline, end of hemodynamic monitoring (about Day 10)
  CPO measured by pulmonary artery catheter

SECONDARY OUTCOMES:
RV failure defined by the 2014 Interagency Registry for Mechanical Circulatory Support (INTERMACS) | Through duration of hospitalization, up to 30 days following LVAD implantation
  The INTERMACS definition of RVF stratifies patients based on duration of inotropic therapy, inhaled nitric oxide therapy, vasodilator therapy or RVAD implantation. RVF is described as mild, moderate, severe, or severe acute based on ≤7, 8-14, >14 days of the above therapies or RVAD implantation, respectively
RV failure defined by the 2020 Academic Research Consortium (ARC) | Through duration of hospitalization, up to 30 days following LVAD implantation
  The ARC definition of RVF stratifies patients based on the onset of RVF (e.g. early acute right heart failure, early post-implant right heart failure, or late right heart failure) requiring inotropic therapy or RVAD implantation during LVAD implantation, <30 days post-operatively, or >30 days post-operatively, respectively
Inotropic therapy | Through duration of hospitalization, up to 30 days following LVAD implantation
  Total number of inotropes used
Vasopressor therapy | Through duration of hospitalization, up to 30 days following LVAD implantation
  Total number of vasopressors used
Total time on inhaled nitric oxide | Through duration of hospitalization, up to 30 days following LVAD implantation
  Measured in days
Number of individuals who experience all-cause mortality | Through duration of hospitalization, up to 30 days following LVAD implantation
  All-cause mortality
ICU length of stay | Through duration of hospitalization, up to 30 days following LVAD implantation
  Measured in days
Hospital length of stay | Through duration of hospitalization, up to 30 days following LVAD implantation
  Measured in days
Number of individuals with acute kidney injuries requiring renal replacement therapy | Through duration of hospitalization, up to 30 days following LVAD implantation
  Acute kidney injury requiring renal replacement therapy (intermittent hemodialysis or continuous renal replacement therapy)
Number of individuals with transient ischemic attacks [TIA] or cerebrovascular accidents [CVA] | Through duration of hospitalization, up to 30 days following LVAD implantation
  Transient ischemic attack or cerebrovascular accident as diagnosed by a Neurologist either clinically and/or radiographically
Number of individuals with an arrhythmia requiring medical team intervention | Through duration of hospitalization, up to 30 days following LVAD implantation
  Arrhythmia requiring medical team intervention, either through electrical or chemical cardioversion or any intravenous anti-arrhythmia medication administration
Number of individuals who need tracheostomy | Through duration of hospitalization, up to 30 days following LVAD implantation
  Need for tracheostomy
Number of individuals needing percutaneous endoscopic gastrostomy tube | Through duration of hospitalization, up to 30 days following LVAD implantation
  Need for percutaneous endoscopic gastrostomy tube

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grinstein, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No